CLINICAL TRIAL: NCT07213999
Title: Evaluating and Understanding the Effects of Deep Brain Stimulation Using Novel Electrophysiology Technique and Device in Parkinson's Disease
Brief Title: Novel DBS Device in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005478; R21NS111214-01 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease (PD)
Keywords: DBS; Deep brain stimulation; Parkinson's disease; PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neural recorder (Experimental)
  Interventions: Device: Novel neural recorder

INTERVENTIONS:
Device: Novel neural recorder — The neural recorder does not suffer saturation from stimulation artifacts, allowing circuits to record neural signals with higher precision.

SUMMARY:
The purpose of this research is to test a new recorder that can measure brain activity when stimulation is turned on during deep brain stimulation (DBS) surgery. To continue to improve DBS therapy, the investigators need to better understand the changes in the brain of people with Parkinson's disease (PD). They also need to know how this is affected by DBS. Current recorders measure activity immediately after, but not during, stimulation. Standard-of-care DBS already includes the electrical recording of brain activity during movement of arms and legs. These recordings occur during the microelectrode recording part of the surgery and are used by the medical team to determine where to place the DBS electrode.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is shown to be very effective in alleviating the motor symptoms of Parkinson's disease (PD). However, its exact mechanism is not well-understood. Clinical studies have reported conflicting results regarding the effects of DBS, with some studies suggesting that it inhibits target neurons while some others suggest that it excites those neurons. One of the significant hurdles plaguing the study of DBS is the large artifacts caused by electrical stimulation. The large artifacts saturate the neural recorder and also make it take a long time to recover to its normal working conditions. Consequently, no reliable neural feedback can be recorded during the high frequency stimulation of DBS. The investigators have developed a new neural recorder that does not saturate even in the presence of large artifacts. The recorder has been validated in animal studies and recently in human experiments. The investigators propose to further develop the device to study the mechanisms of DBS: in Aim 1, they will develop an artifact-resilient neural recorder and related software suite to support intraoperative monitoring during DBS. In Aim 2, they will use the proposed device to carry out an intraoperative electrophysiological recording of the subthalamic nucleus (STN) or globus pallidus internus (GPi) in PD patients. The investigators will compare activities of the neurons when high or low stimulation frequency is used, when stimulation is delivered ipsilaterally or contralaterally, and when different temporal patterns of DBS pulses are used. Measurements of therapeutic effects in terms of tremor power will be obtained by a wireless inertial measurement unit. The investigators will correlate tremor power, neural responses, and stimulation parameters during DBS, which can provide new insights into the mechanisms of DBS. These insights can potentially lead to a better stimulation paradigm that can enhance the efficacy of DBS.

ELIGIBILITY:
Inclusion Criteria:

* Has unilateral STN or GPi DBS and is approved to undergo second or contralateral side implantation;
* Diagnosis of idiopathic PD;
* A history of a good response to levodopa (carbidopa/levodopa) defined as at least a 30% improvement in motor unified Parkinson's disease rating scale (UPDRS) score;
* DBS surgery at UMN is planned as part of routine clinical care.

Exclusion Criteria:

* Other significant neurological disorder
* History of dementia
* Patients with post-operative complications or adverse effects (e.g. ON stimulation dystonias) that affect patient safety or confound the experiment will be excluded from further study
* Pregnant women

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Wireless 9-axis inertial measurement unit (IMU) with 3-axis accelerometer, gyroscope, and magnetometer will quantitatively measure the activity of neurons when high or low stimulation frequency is used. | For the duration of the participant's' DBS surgery.
  The investigators will compare the activity of neurons when high or low stimulation frequency is used, when stimulation is delivered ipsilaterally or contralaterally, and when different temporal patterns of DBS pulses are used within the constraints of standard clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tabbal SD, Ushe M, Mink JW, Revilla FJ, Wernle AR, Hong M, Karimi M, Perlmutter JS. Unilateral subthalamic nucleus stimulation has a measurable ipsilateral effect on rigidity and bradykinesia in Parkinson disease. Exp Neurol. 2008 May;211(1):234-42. doi: 10.1016/j.expneurol.2008.01.024. Epub 2008 Feb 14. PMID 18329019
- [Background] Nakamura K, Christine CW, Starr PA, Marks WJ Jr. Effects of unilateral subthalamic and pallidal deep brain stimulation on fine motor functions in Parkinson's disease. Mov Disord. 2007 Apr 15;22(5):619-26. doi: 10.1002/mds.21300. PMID 17230483
- [Background] Alberts JL, Okun MS, Vitek JL. The persistent effects of unilateral pallidal and subthalamic deep brain stimulation on force control in advanced Parkinson's patients. Parkinsonism Relat Disord. 2008 Aug;14(6):481-8. doi: 10.1016/j.parkreldis.2007.11.014. Epub 2008 Mar 14. PMID 18342565
- [Background] Pogosyan A, Yoshida F, Chen CC, Martinez-Torres I, Foltynie T, Limousin P, Zrinzo L, Hariz MI, Brown P. Parkinsonian impairment correlates with spatially extensive subthalamic oscillatory synchronization. Neuroscience. 2010 Nov 24;171(1):245-57. doi: 10.1016/j.neuroscience.2010.08.068. Epub 2010 Sep 9. PMID 20832452
- [Background] A Low-Noise, Wireless, Frequency-Shaping based Neural Recorder
- [Background] Zhi Yang, Jian Xu, Anh Tuan Nguyen, Tong Wu, Wenfeng Zhao, Wing-Kin Tam. Neuronix enables continuous, simultaneous neural recording and electrical microstimulation. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:4451-4454. doi: 10.1109/EMBC.2016.7591715. PMID 28269266
- [Background] Sharpee TO, Destexhe A, Kawato M, Sekulic V, Skinner FK, Wojcik DK, Chintaluri C, Cserpan D, Somogyvari Z, Kim JK, Kilpatrick ZP, Bennett MR, Josic K, Elices I, Arroyo D, Levi R, Rodriguez FB, Varona P, Hwang E, Kim B, Han HB, Kim T, McKenna JT, Brown RE, McCarley RW, Choi JH, Rankin J, Popp PO, Rinzel J, Tabas A, Rupp A, Balaguer-Ballester E, Maturana MI, Grayden DB, Cloherty SL, Kameneva T, Ibbotson MR, Meffin H, Koren V, Lochmann T, Dragoi V, Obermayer K, Psarrou M, Schilstra M, Davey N, Torben-Nielsen B, Steuber V, Ju H, Yu J, Hines ML, Chen L, Yu Y, Kim J, Leahy W, Shlizerman E, Birgiolas J, Gerkin RC, Crook SM, Viriyopase A, Memmesheimer RM, Gielen S, Dabaghian Y, DeVito J, Perotti L, Kim AJ, Fenk LM, Cheng C, Maimon G, Zhao C, Widmer Y, Sprecher S, Senn W, Halnes G, Maki-Marttunen T, Keller D, Pettersen KH, Andreassen OA, Einevoll GT, Yamada Y, Steyn-Ross ML, Alistair Steyn-Ross D, Mejias JF, Murray JD, Kennedy H, Wang XJ, Kruscha A, Grewe J, Benda J, Lindner B, Badel L, Ohta K, Tsuchimoto Y, Kazama H, Kahng B, Tam ND, Pollonini L, Zouridakis G, Soh J, Kim D, Yoo M, Palmer SE, Culmone V, Bojak I, Ferrario A, Merrison-Hort R, Borisyuk R, Kim CS, Tezuka T, Joo P, Rho YA, Burton SD, Bard Ermentrout G, Jeong J, Urban NN, Marsalek P, Kim HH, Moon SH, Lee DW, Lee SB, Lee JY, Molkov YI, Hamade K, Teka W, Barnett WH, Kim T, Markin S, Rybak IA, Forro C, Dermutz H, Demko L, Voros J, Babichev A, Huang H, Verduzco-Flores S, Dos Santos F, Andras P, Metzner C, Schweikard A, Zurowski B, Roach JP, Sander LM, Zochowski MR, Skilling QM, Ognjanovski N, Aton SJ, Zochowski M, Wang SJ, Ouyang G, Guang J, Zhang M, Michael Wong KY, Zhou C, Robinson PA, Sanz-Leon P, Drysdale PM, Fung F, Abeysuriya RG, Rennie CJ, Zhao X, Choe Y, Yang HF, Mi Y, Lin X, Wu S, Liedtke J, Schottdorf M, Wolf F, Yamamura Y, Wickens JR, Rumbell T, Ramsey J, Reyes A, Draguljic D, Hof PR, Luebke J, Weaver CM, He H, Yang X, Ma H, Xu Z, Wang Y, Baek K, Morris LS, Kundu P, Voon V, Agnes EJ, Vogels TP, Podlaski WF, Giese M, Kuravi P, Vogels R, Seeholzer A, Podlaski W, Ranjan R, Vogels T, Torres JJ, Baroni F, Latorre R, Gips B, Lowet E, Roberts MJ, de Weerd P, Jensen O, van der Eerden J, Goodarzinick A, Niry MD, Valizadeh A, Pariz A, Parsi SS, Warburton JM, Marucci L, Tamagnini F, Brown J, Tsaneva-Atanasova K, Kleberg FI, Triesch J, Moezzi B, Iannella N, Schaworonkow N, Plogmacher L, Goldsworthy MR, Hordacre B, McDonnell MD, Ridding MC, Zapotocky M, Smit D, Fouquet C, Trembleau A, Dasgupta S, Nishikawa I, Aihara K, Toyoizumi T, Robb DT, Mellen N, Toporikova N, Tang R, Tang YY, Liang G, Kiser SA, Howard JH Jr, Goncharenko J, Voronenko SO, Ahamed T, Stephens G, Yger P, Lefebvre B, Spampinato GLB, Esposito E, et Olivier Marre MS, Choi H, Song MH, Chung S, Lee DD, Sompolinsky H, Phillips RS, Smith J, Chatzikalymniou AP, Ferguson K, Alex Cayco Gajic N, Clopath C, Angus Silver R, Gleeson P, Marin B, Sadeh S, Quintana A, Cantarelli M, Dura-Bernal S, Lytton WW, Davison A, Li L, Zhang W, Wang D, Song Y, Park S, Choi I, Shin HS, Choi H, Pasupathy A, Shea-Brown E, Huh D, Sejnowski TJ, Vogt SM, Kumar A, Schmidt R, Van Wert S, Schiff SJ, Veale R, Scheutz M, Lee SW, Gallinaro J, Rotter S, Rubchinsky LL, Cheung CC, Ratnadurai-Giridharan S, Shomali SR, Ahmadabadi MN, Shimazaki H, Nader Rasuli S, Zhao X, Rasch MJ, Wilting J, Priesemann V, Levina A, Rudelt L, Lizier JT, Spinney RE, Rubinov M, Wibral M, Bak JH, Pillow J, Zaho Y, Park IM, Kang J, Park HJ, Jang J, Paik SB, Choi W, Lee C, Song M, Lee H, Park Y, Yilmaz E, Baysal V, Ozer M, Saska D, Nowotny T, Chan HK, Diamond A, Herrmann CS, Murray MM, Ionta S, Hutt A, Lefebvre J, Weidel P, Duarte R, Morrison A, Lee JH, Iyer R, Mihalas S, Koch C, Petrovici MA, Leng L, Breitwieser O, Stockel D, Bytschok I, Martel R, Bill J, Schemmel J, Meier K, Esler TB, Burkitt AN, Kerr RR, Tahayori B, Nolte M, Reimann MW, Muller E, Markram H, Parziale A, Senatore R, Marcelli A, Skiker K, Maouene M, Neymotin SA, Seidenstein A, Lakatos P, Sanger TD, Menzies RJ, McLauchlan C, van Albada SJ, Kedziora DJ, Neymotin S, Kerr CC, Suter BA, Shepherd GMG, Ryu J, Lee SH, Lee J, Lee HJ, Lim D, Wang J, Lee H, Jung N, Anh Quang L, Maeng SE, Lee TH, Lee JW, Park CH, Ahn S, Moon J, Choi YS, Kim J, Jun SB, Lee S, Lee HW, Jo S, Jun E, Yu S, Goetze F, Lai PY, Kim S, Kwag J, Jang HJ, Filipovic M, Reig R, Aertsen A, Silberberg G, Bachmann C, Buttler S, Jacobs H, Dillen K, Fink GR, Kukolja J, Kepple D, Giaffar H, Rinberg D, Shea S, Koulakov A, Bahuguna J, Tetzlaff T, Kotaleski JH, Kunze T, Peterson A, Knosche T, Kim M, Kim H, Park JS, Yeon JW, Kim SP, Kang JH, Lee C, Spiegler A, Petkoski S, Palva MJ, Jirsa VK, Saggio ML, Siep SF, Stacey WC, Bernar C, Choung OH, Jeong Y, Lee YI, Kim SH, Jeong M, Lee J, Kwon J, Kralik JD, Jahng J, Hwang DU, Kwon JH, Park SM, Kim S, Kim H, Kim PS, Yoon S, Lim S, Park C, Miller T, Clements K, Ahn S, Ji EH, Issa FA, Baek J, Oba S, Yoshimoto J, Doya K, Ishii S, Mosqueiro TS, Strube-Bloss MF, Smith B, Huerta R, Hadrava M, Hlinka J, Bos H, Helias M, Welzig CM, Harper ZJ, Kim WS, Shin IS, Baek HM, Han SK, Richter R, Vitay J, Beuth F, Hamker FH, Toppin K, Guo Y, Graham BP, Kale PJ, Gollo LL, Stern M, Abbott LF, Fedorov LA, Giese MA, Ardestani MH, Faraji MJ, Preuschoff K, Gerstner W, van Gendt MJ, Briaire JJ, Kalkman RK, Frijns JHM, Lee WH, Frangou S, Fulcher BD, Tran PHP, Fornito A, Gliske SV, Lim E, Holman KA, Fink CG, Kim JS, Mu S, Briggman KL, Sebastian Seung H; the EyeWirers; Wegener D, Bohnenkamp L, Ernst UA, Devor A, Dale AM, Lines GT, Edwards A, Tveito A, Hagen E, Senk J, Diesmann M, Schmidt M, Bakker R, Shen K, Bezgin G, Hilgetag CC, van Albada SJ, Sun H, Sourina O, Huang GB, Klanner F, Denk C, Glomb K, Ponce-Alvarez A, Gilson M, Ritter P, Deco G, Witek MAG, Clarke EF, Hansen M, Wallentin M, Kringelbach ML, Vuust P, Klingbeil G, De Schutter E, Chen W, Zang Y, Hong S, Takashima A, Zamora C, Gallimore AR, Goldschmidt D, Manoonpong P, Karoly PJ, Freestone DR, Soundry D, Kuhlmann L, Paninski L, Cook M, Lee J, Fishman YI, Cohen YE, Roberts JA, Cocchi L, Sweeney Y, Lee S, Jung WS, Kim Y, Jung Y, Song YK, Chavane F, Soman K, Muralidharan V, Srinivasa Chakravarthy V, Shivkumar S, Mandali A, Pragathi Priyadharsini B, Mehta H, Davey CE, Brinkman BAW, Kekona T, Rieke F, Buice M, De Pitta M, Berry H, Brunel N, Breakspear M, Marsat G, Drew J, Chapman PD, Daly KC, Bradle SP, Seo SB, Su J, Kavalali ET, Blackwell J, Shiau L, Buhry L, Basnayake K, Lee SH, Levy BA, Baker CI, Leleu T, Philips RT, Chhabria K. 25th Annual Computational Neuroscience Meeting: CNS-2016. BMC Neurosci. 2016 Aug 18;17 Suppl 1(Suppl 1):54. doi: 10.1186/s12868-016-0283-6. PMID 27534393
- [Background] Xu J, Wu T, Liu W, Yang Z. A frequency shaping neural recorder with 3 pF input capacitance and 11 plus 4.5 bits dynamic range. IEEE Trans Biomed Circuits Syst. 2014 Aug;8(4):510-27. doi: 10.1109/TBCAS.2013.2293821. PMID 25073127
- [Background] Baker KB, Zhang J, Vitek JL. Pallidal stimulation: effect of pattern and rate on bradykinesia in the non-human primate model of Parkinson's disease. Exp Neurol. 2011 Oct;231(2):309-13. doi: 10.1016/j.expneurol.2011.06.012. Epub 2011 Jul 1. PMID 21767534
- [Background] Birdno MJ, Kuncel AM, Dorval AD, Turner DA, Grill WM. Tremor varies as a function of the temporal regularity of deep brain stimulation. Neuroreport. 2008 Mar 26;19(5):599-602. doi: 10.1097/WNR.0b013e3282f9e45e. PMID 18388746
- [Background] Dorval AD, Kuncel AM, Birdno MJ, Turner DA, Grill WM. Deep brain stimulation alleviates parkinsonian bradykinesia by regularizing pallidal activity. J Neurophysiol. 2010 Aug;104(2):911-21. doi: 10.1152/jn.00103.2010. Epub 2010 May 26. PMID 20505125
- [Background] Johnson LA, Nebeck SD, Muralidharan A, Johnson MD, Baker KB, Vitek JL. Closed-Loop Deep Brain Stimulation Effects on Parkinsonian Motor Symptoms in a Non-Human Primate - Is Beta Enough? Brain Stimul. 2016 Nov-Dec;9(6):892-896. doi: 10.1016/j.brs.2016.06.051. Epub 2016 Jun 22. PMID 27401045
- [Background] Hess CW, Vaillancourt DE, Okun MS. The temporal pattern of stimulation may be important to the mechanism of deep brain stimulation. Exp Neurol. 2013 Sep;247:296-302. doi: 10.1016/j.expneurol.2013.02.001. Epub 2013 Feb 8. PMID 23399890
- [Background] 15-DOF motor decoding based on a high performance PNS interface and deep neural network
- [Background] Galati S, Mazzone P, Fedele E, Pisani A, Peppe A, Pierantozzi M, Brusa L, Tropepi D, Moschella V, Raiteri M, Stanzione P, Bernardi G, Stefani A. Biochemical and electrophysiological changes of substantia nigra pars reticulata driven by subthalamic stimulation in patients with Parkinson's disease. Eur J Neurosci. 2006 Jun;23(11):2923-8. doi: 10.1111/j.1460-9568.2006.04816.x. PMID 16819981
- [Background] Lafreniere-Roula M, Kim E, Hutchison WD, Lozano AM, Hodaie M, Dostrovsky JO. High-frequency microstimulation in human globus pallidus and substantia nigra. Exp Brain Res. 2010 Aug;205(2):251-61. doi: 10.1007/s00221-010-2362-8. Epub 2010 Jul 17. PMID 20640411
- [Background] Dostrovsky JO, Levy R, Wu JP, Hutchison WD, Tasker RR, Lozano AM. Microstimulation-induced inhibition of neuronal firing in human globus pallidus. J Neurophysiol. 2000 Jul;84(1):570-4. doi: 10.1152/jn.2000.84.1.570. PMID 10899228
- [Background] Beurrier C, Bioulac B, Audin J, Hammond C. High-frequency stimulation produces a transient blockade of voltage-gated currents in subthalamic neurons. J Neurophysiol. 2001 Apr;85(4):1351-6. doi: 10.1152/jn.2001.85.4.1351. PMID 11287459
- [Background] Tai CH, Boraud T, Bezard E, Bioulac B, Gross C, Benazzouz A. Electrophysiological and metabolic evidence that high-frequency stimulation of the subthalamic nucleus bridles neuronal activity in the subthalamic nucleus and the substantia nigra reticulata. FASEB J. 2003 Oct;17(13):1820-30. doi: 10.1096/fj.03-0163com. PMID 14519661
- [Background] Toleikis JR, Metman LV, Pilitsis JG, Barborica A, Toleikis SC, Bakay RA. Effect of intraoperative subthalamic nucleus DBS on human single-unit activity in the ipsilateral and contralateral subthalamic nucleus. J Neurosurg. 2012 May;116(5):1134-43. doi: 10.3171/2011.12.JNS102176. Epub 2012 Feb 17. PMID 22339160
- [Background] Filali M, Hutchison WD, Palter VN, Lozano AM, Dostrovsky JO. Stimulation-induced inhibition of neuronal firing in human subthalamic nucleus. Exp Brain Res. 2004 Jun;156(3):274-81. doi: 10.1007/s00221-003-1784-y. Epub 2004 Jan 24. PMID 14745464
- See also: Related Info — https://reporter.nih.gov/project-details/9722638